CLINICAL TRIAL: NCT01919216
Title: Placebo Effects in the Treatment of Depression: Cognitive and Neural Mechanisms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bret Rutherford, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6038/6996R; K23MH085236 (NIH)
Record Dates: First submitted 2013-08-05; First posted 2013-08-08 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Open Track (Active Comparator): Open treatment with 20mg of citalopram, increased to 40mg if depression has not remitted at week 4.
  Interventions: Drug: Citalopram
- Placebo Track (Placebo Comparator): Blinded treatment with either citalopram 20mg or placebo, increased to citalopram 40mg or placebo at week 4 if depression has not remitted.
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Citalopram
  Other Names: Celexa

SUMMARY:
Studies of the neural mechanisms underlying placebo effects in antidepressant clinical trials largely have been limited to demonstrating objective differences in brain activity between responders and non-responders to placebo. This 8 week Placebo-controlled and Open groups study employs a novel antidepressant trial design with integrated functional magnetic resonance imaging (fMRI) to manipulate patient expectancy and examine its neural mediators.

DETAILED DESCRIPTION:
The placebo effect represents a potent treatment for Major Depressive Disorder (MDD)-placebo response in acute randomized controlled trials (RCTs) of antidepressant medications averages 30%, and meta-analyses have estimated the proportion of medication response attributable to placebo to be 50-75%. Patient expectancy is the mechanism of placebo effects in antidepressant RCTs and has been positively associated with medication response. Determining how expectancy alters the course of MDD could lead to methods of optimizing placebo effects and improving the treatment of MDD. In addition, investigating the neurobiology of placebo effects has the potential to elucidate the pathophysiology of MDD and the mechanisms of action of antidepressant treatments. Brain regions implicated in expectancy and placebo effects comprise prefrontal cortical (PFC) areas, amygdala, insular cortex, rostral anterior cingulate cortex (rACC), and dopaminergic reward pathways in the striatum. Pathological decreases in PFC and striatal function, increases in limbic activity, and disordered connectivity between these regions have all been observed in MDD, and the rostral and dorsal ACC have been repeatedly linked to antidepressant treatment response.

Therefore, studying placebo effects offers a window into the functioning of the neural circuits that are disturbed in MDD and improve with effective treatment. The goals of this study are to determine whether expectancy affects the outcome of antidepressant pharmacotherapy and to investigate the neural mechanisms of expectancy effects. These will be accomplished by conducting a clinical trial randomizing adult outpatients with MDD to 8 weeks of treatment in high vs. low expectancy conditions. The high expectancy condition will be open administration of citalopram, while the low expectancy condition will be placebo-controlled administration of citalopram. The neural mechanisms of expectancy will be determined using functional Magnetic Resonance Imaging (fMRI) paradigms to investigate treatment activation differences in brain regions associated with placebo effects and MDD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 24-75 years
* Diagnosed with Diagnostic and Statistical Manual of Mental Disorders (DSM) IV Major Depressive Disorder, nonpsychotic
* 24-item Hamilton Rating Scale for Depression (HRSD) score ≥ 16
* Willing to and capable of providing informed consent and complying with study procedures
* Subjects are right-handed
* Using appropriate contraceptive method if woman of child-bearing age

Exclusion Criteria:

* Current comorbid Axis I DSM IV disorder other than Nicotine Dependence, Adjustment Disorder, Panic Disorder, Generalized Anxiety Disorder, or Social Phobia
* Diagnosis of substance abuse or dependence (excluding Nicotine Dependence) within the past 12 months
* History of psychosis or psychotic disorder, mania or bipolar disorder
* Subject is considered to be at significant risk of suicide based on current mental status and recent history
* History of allergic or adverse reaction to citalopram, or nonresponse to adequate trial of citalopram (at least 4 weeks at dose of 40mg) or escitalopram (at least 4 weeks at dose of 20mg)
* Subject is considered based on history to be unlikely to respond to the single agent citalopram (i.e., subjects with treatment resistant depression)
* Current treatment with psychotherapy
* Clinical Global Impression (CGI)-Severity score of 7 at baseline Clinical Interview
* Current or recent (within the past 4 weeks) treatment with any of the following: antidepressants, antipsychotics, mood stabilizers, isoniazid, glucocorticoids, opiates, centrally active antihypertensive drugs (e.g. clonidine, reserpine)
* Subject has metal in body or prior history working with metal fragments (e.g., as a machinist), tattoos, or unable to tolerate the scanning procedures (i.e., severe obesity, claustrophobia)
* Acute, severe, or unstable medical illness

Ages: 24 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret R Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Rutherford BR, Roose SP. A model of placebo response in antidepressant clinical trials. Am J Psychiatry. 2013 Jul;170(7):723-33. doi: 10.1176/appi.ajp.2012.12040474. PMID 23318413
- [Derived] Zilcha-Mano S, Wang Z, Peterson BS, Wall MM, Chen Y, Wager TD, Brown PJ, Roose SP, Rutherford BR. Neural mechanisms of expectancy-based placebo effects in antidepressant clinical trials. J Psychiatr Res. 2019 Sep;116:19-25. doi: 10.1016/j.jpsychires.2019.05.023. Epub 2019 May 26. PMID 31176108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the Adult and Late Life Depression Research Clinic at the New York State Psychiatric Institute (NYSPI) and approved by the NYSPI Institutional Review Board. Recruitment period started January 2010 and ended in June 2016.
Pre-assignment Details: 11 enrolled participants were lost to follow up prior to randomization.
Groups:
- Open Track: Open treatment with 20mg of citalopram, increased to 40mg if depression has not remitted at week 4.
  Citalopram
- Placebo Track - Citalopram: Blinded treatment with either citalopram 20mg, increased to citalopram 40mg at week 4 if depression has not remitted.
  Citalopram
- Placebo Track - Placebo: Blinded treatment with either placebo
Period: Overall Study
Arm/Group | Open Track | Placebo Track - Citalopram | Placebo Track - Placebo
Started | 28 | 21 | 5
Completed | 26 | 20 | 4
Not Completed | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Track - Citalopram: Blinded treatment with citalopram 20mg , increased to citalopram 40mg at week 4 if depression has not remitted.
  Citalopram
- Placebo Track - Placebo: Blinded treatment with placebo
- Total: Total of all reporting groups
Arm/Group | Open Track | Placebo Track - Citalopram | Placebo Track - Placebo | Total
Number analyzed (Participants) | 26 | 20 | 4 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 20 | 4 | 50
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12) | 43.8 (10.7) | 34.3 (10.2) | 41.79 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 3 | 30
  Male | 9 | 10 | 1 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 1 | 8
  Not Hispanic or Latino | 21 | 18 | 3 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 1 | 14
  White | 12 | 13 | 3 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 20 | 4 | 50
Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — The patient is rated by a clinician among 24 dimensions with a score on a 3 or 5 point scale. A score of 0-9 is considered to be normal. Score between 10-18 is considered as mild depression, Scores between 19-26 indicate moderate, scores between 27-34 indicate severe, and score between 35-75 indicate very severe depression.
  units on a scale | 25.7 (5.5) | 25.7 (4.1) | 23.8 (2.8) | 25.55 (4.8)
Hamilton Anxiety Rating Scale (HAM-A) [Mean (Standard Deviation); unit: units on a scale] — HAM-A consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe). The summation of each of the 14 individually rated items will yield a comprehensive score in the range of 0 to 56. It has been predetermined that the results of the evaluation can be interpreted as follows. A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity. Lastly, a score of 25 to 30 indicates a moderate to severe anxiety severity.
  units on a scale | 13.2 (4.9) | 15.1 (4.8) | 16.7 (9.2) | 14.24 (5.34)
CGI Severity [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment: 0 normal, not at all ill to 7 Among the most extremely ill patients
  units on a scale | 4.4 (0.6) | 4.3 (0.5) | 4.3 (0.6) | 4.35 (0.56)
Quick Inventory of Depressive Symptoms-Self Report (QIDS-SR) 16 Item Scale [Mean (Standard Deviation); unit: units on a scale] — The16 item Quick Inventory of Depressive Symptomatology (QIDS) contains 16 questions score from 0 to 3 each.
  Qids score 1-5, not depressed; 6-10, Mild depression; 11-15, Moderate depression; 16-20, Severe depression; 21-27, very severe depression
  units on a scale | 19.7 (5.2) | 19.8 (7.2) | 17.8 (7.5) | 19.59 (6.27)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression
Description: The patient is rated by a clinician among 24 dimensions with a score on a 3 or 5 point scale. A score of 0-9 is considered to be normal. Score between 10-18 is considered as mild depression, Scores between 19-26 indicate moderate, scores between 27-34 indicate severe, and score between 35-75 indicate very severe depression.
Time Frame: 8 weeks
Population: 54 subjects participated in the study, of whom 4 (2 in open track, 1 in placebo track - citalopram, 1 in placebo track - placebo) were lost to follow-up prior to taking the study medication and were excluded from the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Track - Citalopram: Blinded treatment with either citalopram 20mg, increased to citalopram 40mg or placebo at week 4 if depression has not remitted.
  Citalopram
Arm/Group | Open Track | Placebo Track - Citalopram | Placebo Track - Placebo
Number analyzed (Participants) | 26 | 20 | 4
units on a scale | 10.79 (8.96) | 15.30 (9.2) | 12.75 (5.188)

ADVERSE EVENTS:
Groups:
- Placebo Track - Citalopram: Blinded treatment with citalopram 20mg, increased to citalopram 40mg or placebo at week 4 if depression has not remitted.
  Citalopram
Arm/Group | Open Track | Placebo Track - Citalopram | Placebo Track - Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/20 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/20 | 0/4
Other Adverse Events (participants affected / at risk) | 0/26 | 0/20 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No